CLINICAL TRIAL: NCT05480293
Title: A Phase III, Multicenter, Randomized, Double-Masked, Parallel Controlled, Non Inferior Study to Compare the Efficacy and Safety of SCT510A Administered by Intravitreal Injection With Ranibizumab in Subjects With Wet Age-related Macular Degeneration (wAMD)
Brief Title: This Study Will Compare the Efficacy and Safety of SCT510A Administered by Intravitreal Injection (IVT) With Ranibizumab in Patients With wAMD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCT510A-A301
Record Dates: First submitted 2022-07-28; First posted 2022-07-29 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-05

CONDITIONS: Wet Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCT510A (Experimental): SCT510A(1.25mg), Vitreous injection, injection once every 4 weeks
  Interventions: Drug: SCT510A
- Ranibizumab (Active Comparator): Ranibizumab(0.5mg), Vitreous injection, injection once every 4 weeks
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — ranibizumab，0.5mg,IVT
  Arms: Ranibizumab
Drug: SCT510A — SCT510A，1.25mg,IVT
  Arms: SCT510A

SUMMARY:
The purpose of this study is to compare the efficacy and safety of SCT510A versus Lucentis in the treatment of wet age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form;
2. Age≥45 years，male or femal;
3. The study eye must meet the following criteria： Diagnosis of wAMD； Primary or recurrent active subfoveal or parafoveal choroidal neovascularization (CNV) lesions secondary to wAMD； The total lesion area ≤ 30mm2； The BCVA letters between 19 and 73, inclusive, in the study eye, using Early Treatment Diabetic Retinopathy Study (ETDRS) charts；
4. The study eye has not received any anti-VEGF treatment within 3 months before randomization, such as ranibizumab, bevacizumab, conbercept, etc；

Exclusion Criteria:

1. Macular-related retinal pigment epithelial tears in the study eye; scar, fibrosis, atrophy or dense subfoveal exudation involving the fovea in the study eye;
2. Significant afferent pupillary defect (APD) in the study eye；
3. Aphakia (except intraocular lens) or posterior capsular rupture of the lens (except yttrium aluminium-garnet (YAG) laser posterior capsulotomy after intraocular lens implantation ≥1 month before randomization) in the study eye.
4. The study eye has any eye diseases or medical history other than nAMD that may affect central vision and/or macular examine (diabetic retinopathy, retinal vein occlusion, retinal detachment, macular hole, macular epiretinal membrane, vitreous macular traction syndrome, optic nerve disease, etc.);
5. CNV caused by non-nAMD exists in the study eye (such as trauma, ocular histoplasmosis, vascular stripes, etc.);
6. The study eye has high myopia with diopter≥8D;
7. The study eye has poorly controlled glaucoma (defined as intraocular pressure≥25 mmHg after anti-glaucoma treatment), or has received glaucoma filtering surgery;
8. Vitreous hemorrhage in the study eye before randomization;
9. Any history of the following ophthalmic surgery in the study eye: vitrectomy, macular transposition; any evidence of external eye surgery within 1 month, cataract surgery within 2 months or other intraocular surgery within 3 months before randomization in the study eye;
10. Active inflammation or infection in either eye, such as conjunctivitis,keratitis, scleritis, or endophthalmitis, ect；
11. Previous IVT injection of any anti-VEGF drug into fellow eye within 3 months before randomization;
12. Fellow eye uses ETDRS testing to detect BCVA <19 letters;
13. Known allergy to any component of the study intervention or history of allergy to fluorescein or indocyanine green, any anesthetics or antimicrobial agents used during the course of the study;
14. Abnormal liver and kidney function (ALT, AST≥2.5 times the upper limit of normal; total bilirubin≥1.5 times the upper limit of normal; serum creatinine≥1.5 times the upper limit of normal);Abnormal coagulation function（prothrombin time ≥ 3 seconds over ULN, activated partial thromboplastin time ≥ 10 seconds over ULN）;
15. Poorly-controlled blood pressure (defined as: after receiving antihypertensive drugs, the subject's systolic value ≥160 mmHg or diastolic value ≥100 mmHg at seat);
16. History of a medical condition, including myocardial infarction, unstable angina pectoris, cerebrovascular accidents (including TIA), other thromboembolic diseases (such as thromboembolic angiitis, pulmonary embolism, deep vein thrombosis, portal vein thrombosis, etc.) within 6 months before randomization;
17. Any history of surgery within 1 month before randomization, and/or any currently unhealed wounds, ulcers, fractures, etc.;
18. Evidence of significant uncontrolled concomitant diseases such as cardiovascular diseases, nervous system diseases, respiratory system diseases, urinary system diseases, digestive system diseases and endocrine diseases before randomization; uncontrolled diabetes (defined as HbA1c>10.0%);current treatment for active systemic infection;
19. Participated in any drug (other than vitamins and minerals) or device clinical trials within 3 months or the duration of 5 half-lives of the study drug (which is longer) before randomization and have used the test drug or received device treatment.
20. Pregnant, lactating women and the patients who can not take contraceptive measures.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in BCVA at at Week 48 | up to at Week 48
  Change from Baseline in BCVA as measured by Early Treatment Diabetic Retinopathy Study(ETDRS) letter score at week 48.

SECONDARY OUTCOMES:
Proportion of patients gaining at least 5，10，15 letters in the BCVA at Week 12, 24 and 48 | up to Week 12, 24 and 48
  Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.
Mean change from baseline in BCVA at at Week 12 and 24 | up to Week 12 and 24
  Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.
Mean change from baseline in CRT on OCT at Week 12, 24 and 48 (as measured by the Reading Center) | up to Week 12,24 and 48
Mean change from baseline in size of CNV and total area of fluorescein leakage from CNV on FA at Week 12 and 48 (as measured by the Reading Center) | up to Week 12 and 48

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China